CLINICAL TRIAL: NCT04739670
Title: A Single Arm Phase II Trial Evaluating the Efficacy and Safety of Bevacizumab, Carboplatin, Gemcitabine and Atezolizumab in Early Relapsing Metastatic Triple Negative Breast Cancer
Brief Title: Evaluating the Efficacy and Safety of Bevacizumab, Carboplatin, Gemcitabine and Atezolizumab in Breast Cancer
Acronym: BELLA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19/002
Record Dates: First submitted 2021-01-27; First posted 2021-02-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; TNBC; Early relapse; immunotherapy; PD-L1; stromal TILs
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Recurrence | interventions — atezolizumab; Bevacizumab; Gemcitabine; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a multi-center, single arm phase II study designed to evaluate the efficacy and safety of atezolizumab plus bevacizumab plus carboplatin plus gemcitabine in patients with locally recurrent, inoperable or metastatic recurrent PD-L1 positive or stromal TIL positive TNBC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab, Bevacizumab, Gemcitabine and Carboplatin (Experimental): Atezolizumab 1200 mg Day 1 of each 21 day cycle IV, Bevacizumab 15 mg/kg Day 1 of each 21 day cycle IV, Gemcitabine 1000 mg/m2 Day 1 and 8 of each 21 day cycle IV, Carboplatin AUC 5 Day 1 of each 21 day cycle IV
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is a monoclonal antibody of IgG1 isotype PD-L1. It is used across a number of tumour types, both as a single-agent and in combination with other therapies such as chemotherapy.
Drug: Bevacizumab — Bevacizumab is a monoclonal antibody to vascular endothelial growth factor (VEGF) which exerts its effect by inhibiting angiogenesis, a critical component of tumour growth and metastasis.
Drug: Gemcitabine — Gemcitabine is a type of chemotherapy drug
Drug: Carboplatin — Carboplatin is platinum based chemotherapy drug

SUMMARY:
The study hypothesise that the combination of carboplatin, gemcitabine, bevacizumab and atezolizumab may be synergistic and improve outcomes for patients with early relapsed TNBC by overcoming mechanisms of immune resistance and thus potentiating greater and more durable responses to immune checkpoint inhibitor therapy. Early relapsing TNBC represents a high priority, unmet need whereby effective therapeutic strategies are urgently needed.

DETAILED DESCRIPTION:
This is a multi-center, single arm phase II study designed to evaluate the efficacy and safety of atezolizumab plus bevacizumab plus carboplatin plus gemcitabine in patients with locally recurrent, inoperable or metastatic recurrent PD-L1 positive or stromal TIL positive TNBC (Triple Negative Breast Cancer).

Assessment of Programmed death-ligand 1 (PD-L1) status will be available centrally for patients in which PD-L1 testing or stromal TIL testing has not been performed or is not available. In such cases, patients will be required to sign a pre-screening consent form allowing collection and testing of archival tumour samples for PD-L1 status. Patient's that are PD-L1 positive and who fulfil the remaining study eligibility criteria will then be offered participation into the main BELLA study.

Following confirmation of eligibility and registration to the main study, patients will receive treatment as outlined in Table 1 until disease progression according to RECIST 1.1, unacceptable toxicity or patient withdrawal. In the absence of disease progression, the discontinuation of atezolizumab, bevacizumab, carboplatin or gemcitabine (owing to AEs) can occur independently. In the event of ongoing clinical benefit but disease progression, treatment continuation may occur if approved by the CPI.

Table 1:

Order Treatment Dose Dose Frequency Route of Administration

1. Atezolizumab 1200 mg Day 1 of each 21 day cycle IV
2. Bevacizumab 15 mg/kg Day 1 of each 21 day cycle IV
3. Gemcitabine 1000 mg/m2 Day 1 and 8 of each 21 day cycle IV
4. Carboplatin AUC 5 Day 1 of each 21 day cycle IV

Tumour response will be evaluated according to RECIST 1.1. Any evaluable and measurable disease must be documented at screening and re-assessed every 6 weeks from cycle 1 - day 1, regardless of any dose delays.

CT or MRI scans should include chest, abdomen, and pelvis. CT or MRI scans of the brain should be completed at screening and subsequently performed if clinically indicated. At the Investigator's discretion, CT or MRI scans may be repeated at any time if progressive disease is suspected. Imaging based assessments should always be completed rather than clinical assessment to determine response.

Patients who discontinue treatment for any reason will have an End of Treatment visit 30 days after the last dose of treatment after which, patients will move into the follow-up phase of the study where they will be assessed on a 3 monthly basis. Patients with progressive disease will be followed for survival only and patients who discontinue treatment for other reasons will be followed for progression and survival. All patients will be followed up for 2 years after the last patient has been commenced treatment.

There will be 31 patients recruited into the study. If a patient does not receive any protocol treatments for any reason, that patient will be replaced in the study. There are no requirements for follow-up on patients who do not commence treatment.

It is expected that it will take 24 months to accrue the required 31 evaluable patients. Patients will be followed up until 2 years after the last patient has commenced treatment.

Translational Research:

1. Pre-treatment archival FFPE sample collected at pre-screening or screening for the main study will be tested retrospectively at the completion of the trial for

   Quantification of PD-L1 expression and Quantification of TILs on H&E slides
2. Two fresh tumour tissue samples to be collected if deemed clinically feasible by the investigator: an "on-treatment" tumour sample should be collected during cycle 1, days 15-21 and a "post-progression" tumour sample should be collected ≥ 14 days after the last dose of bevacizumab, and prior to commence of a new therapy. On-treatment FFPE sample will be tested for

   Quantification of PD-L1 expression Quantification of TILs on H&E slides
3. A whole blood sample will also be taken prior to the start of treatment, prior to day 1 of cycle 3, and at disease progression (EoT visit) for future research purposes for the assessment of biomarkers of immune activation in peripheral blood mononuclear cells.

Optional biomarker research:

1. If the patient has consented to the Optional Biomarker Study, an additional whole blood sample will be taken on Cycle 1 Day 1 prior starting the treatment for germline whole-genome SNP genotyping to be performed retrospectively.
2. If the patient has consented to the Optional Biomarker Study, stool samples for microbiome analysis will be collected prior to the start of treatment, prior to day 1 of cycle 3, and at disease progression (EoT visit). Microbiome analysis will be performed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Male or female aged 18 years or over
3. Histologically documented triple negative breast cancer (TNBC) that is locally advanced or metastatic and is not amenable to resection with curative intent Receptor status at study entry should correspond to the evaluation of the most recent biopsy as assessed locally TNBC for this study is defined as human epidermal growth factor receptor 2 (HER2)-negative by ASCO-CAP 2018 guidelines, and estrogen receptor (ER) expression < 10%, and progesterone receptor (PgR) expression < 10%
4. PD-L1 positive tumour or tumour-infiltrating lymphocyte-positive defined as:

   Immune cell PD-L1 expression ≥ 1% via SP142 assay via local or central lab OR Stromal TILs ≥ 5% by assessment on H&E stained tumour sections via local laboratory Note: Where possible, local or central testing should be done on the most recently available tumour specimen and must have been obtained within 12 months prior to the date of consent.
5. Documented disease progression (e.g., with biopsy sample, pathology, or imaging report) occurring within 12 months (<12 months) from the last treatment with curative intent, which meets one of the following:

   Date of the last chemotherapy administration or Date of last curative intent adjuvant radiation therapy or Date of the primary breast tumour surgery after neoadjuvant treatment, whichever occurred last
6. Have not received prior chemotherapy or targeted systemic therapy for their locally advanced inoperable or metastatic recurrence Note: Prior radiation therapy for recurrent disease is permitted. There is no required minimum washout period for radiation therapy; however, patients should have recovered from the effects of radiation prior to registration.
7. Measurable disease, as defined by RECIST 1.1 Note: previously irradiated lesions may be considered as measurable disease only if disease progression has been unequivocally documented at that site since radiation.
8. Availability of a representative FFPE tumour block (preferred) or at least 25 unstained slides collected within 12 months prior to registration Note: An FFPE block/slides will not be required for cases where tumour tissue was previously sent to the Central Laboratory for PD-L1 status testing in pre-screening following discussion with the CPI.

   Note: If a tumour sample taken within 12 months before registration is not available and a tumour biopsy is not clinically feasible, the primary surgical resection sample or the most recent FFPE tumour biopsy sample may be used.

   Note: Patients with fewer than 25 unstained slides (but no fewer than 17) may be eligible following discussion with the CPI.
9. Patients with an ECOG performance status 0-1 (see Appendix 1)
10. Life expectancy ≥ 12 weeks
11. Adequate haematologic and end-organ function, defined by the following laboratory results obtained within 7 days prior to registration:

    ANC ≥ 1.5x109/L (without G-CSF support within 2 weeks prior to registration) Lymphocyte count ≥ 0.5x109/L Platelet count ≥ 100x109/L (without transfusion within 2 weeks prior to registration) Haemoglobin ≥ 80 g/L (patients may be transfused or receive erythropoietic treatment to meet this criterion)

    AST and ALT ≤ 2.5 x the ULN, with the following exceptions:
    * Patients with documented liver metastases: AST and ALT ≤ 5× ULN Serum bilirubin ≤ 1.5× ULN
    * Patients with known Gilbert's disease who have serum bilirubin level ≤ 3× ULN may be enrolled.

    Patients who are not receiving therapeutic anticoagulation: INR and aPTT ≤ 1.5× ULN. Patients who are receiving an anticoagulant medicinal product must be on a stable anticoagulant regimen and have an INR which is not above the target therapeutic range during the 7 days prior to registration Calculated CrCl ≥ 30 mL/min (Cockcroft-Gault formula; see Appendix 2).
12. Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of ≤1% per year during the treatment period and for at least 6 months after the last dose of study treatment (see section 7.11.1.1)
13. Women of child bearing potential must have a negative serum pregnancy test within 7 days prior to registration to the study
14. Men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agree to refrain from donating sperm as defined in section 7.11.1.2
15. Patient is willing and able to comply with the protocol for the duration of the study including undergoing biopsies, treatment, and scheduled visits and examination including follow up

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to registration to study
2. Symptomatic, untreated, or actively progressing CNS metastases. Patients with a history of treated CNS lesions are eligible, provided that all of the following criteria are met:

   Measurable or non-measurable disease, per RECIST 1.1, must be present outside the CNS No history of intracranial haemorrhage or spinal cord haemorrhage Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord) There is no clinical or radiological evidence of interim progression between completion of CNS-directed therapy and the screening brain scan The patient has not received stereotactic radiotherapy within 7 days prior to registration to the study or whole-brain radiotherapy within 14 days prior to registration to the study The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan
3. Grade ≥ 2 peripheral neuropathy
4. History or presence of leptomeningeal disease
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) (patients with indwelling catheters such as PleurX® are allowed)
6. Uncontrolled tumour-related pain Note: Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g. bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to registration to the study. Patients should be recovered from the effects of radiation prior to registration. There is no required minimum recovery period. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g. epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco-regional therapy, if appropriate, prior to registration to the study.
7. Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionised calcium or total calcium >3 mmol/L or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy Note: Patients who are receiving bisphosphonate therapy specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcaemia are eligible
8. Malignancies other than TNBC within 5 years prior to registration to the study, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS rate ≥ 90%) and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localised prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer)
9. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to registration, unstable arrhythmias, or unstable angina Note: Patients with a known LVEF < 40% will be excluded Note: Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF 40-50% must be on a stable medical regimen that is optimised in the opinion of the treating physician, in consultation with a cardiologist if appropriate
10. Presence of an abnormal ECG that is clinically significant in the Investigator's opinion, including complete left bundle branch block, second or third-degree heart block, evidence of prior myocardial infarction, or QTcF > 470 ms demonstrated by at least two consecutive ECGs
11. Severe infection requiring oral or IV antibiotics within 4 weeks prior to registration to the study, including but not limited to hospitalisation for complications of infection, bacteraemia, or severe pneumonia Note: patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
12. Positive HIV test at screening
13. Patients with active hepatitis B (chronic or acute; defined as having a positive HBsAg test at screening) or hepatitis C Note: Patients with past HBV infection or resolved HBV infection (defined as the presence of HBc Ab and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to registration Note: Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA
14. Major surgical procedure within 4 weeks prior to registration to the study or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis Note: placement of central venous access catheter(s) (e.g. port or similar) is not considered a major surgical procedure and is therefore permitted
15. Treatment with investigational therapy within 28 days prior to registration
16. Pregnant or lactating, or intending to become pregnant during or within 6 months after the last dose of study treatment
17. Any other significant uncontrolled disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications. This includes significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
18. Poor peripheral venous access
19. Known sensitivity to any component of atezolizumab, bevacizumab, carboplatin and/or gemcitabine Exclusion Criteria Related to Atezolizumab
20. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanised antibodies or fusion proteins
21. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation
22. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, SLE, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with the following are eligible:

    History of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone Controlled Type 1 diabetes mellitus on a stable insulin dosing regimen

    Eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g. patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    Rash must cover less than 10% of body surface area Disease is well controlled prior to registration and only requires low potency topical steroids No acute exacerbations of underlying condition within the previous 12 months (not requiring PUVA, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral steroids)
23. Prior allogeneic stem cell or solid organ transplantation
24. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organising pneumonia (i.e. bronchiolitis obliterans, cryptogenic organising pneumonia), or evidence of active pneumonitis on screening chest CT scan Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
25. Active tuberculosis
26. Receipt of a live, attenuated vaccine within 4 weeks prior to registration or anticipation that a live, attenuated vaccine will be required during atezolizumab treatment or within 5 months after the last dose of atezolizumab
27. Prior treatment with CD137 agonists, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway targeting agents
28. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to registration
29. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, mycophenolate and anti-TNF agents) within 2 weeks prior to registration, or anticipated requirement for systemic immunosuppressive medications during the trial Note: Patients who have received acute, low dose, systemic immunosuppressant medications (e.g. one-time dose of dexamethasone) may be enrolled in the study Note: The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g. fludrocortisone) for patients with orthostatic hypotension, and low dose supplemental corticosteroids (<10 mg prednisone or equivalent) for adrenocortical insufficiency are allowed Exclusion Criteria Related to Bevacizumab
30. Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) Note: Anti-hypertensive therapy to achieve these parameters is allowable
31. Prior history of hypertensive crisis or hypertensive encephalopathy
32. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to registration
33. History of hemoptysis (≥ one-half teaspoon of bright red blood per episode) within 1 month prior to registration
34. Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
35. Current or recent (within 10 days prior to registration) use of aspirin (> 325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and clostazol
36. Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for > 2 weeks prior to registration

    * The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks prior to registration
    * Prophylactic anticoagulation for the patency of venous access devices is allowed
    * Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted. Concomitant treatment with Direct Oral Anticoagulants is not recommended due to bleeding risks
37. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to registration
38. History of abdominal or tracheosphageal fistula or gastrointestinal perforation within 6 months prior to registration
39. Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
40. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
41. Serious, non-healing wound, active ulcer, or untreated bone fracture
42. Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection Note: All patients with ≥ 2+ protein on dipstick urinalysis at screening must undergo a 24-hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Assessed after commencement of treatment, until the last registered patient has been followed up for 2 years.
  PFS is measured from treatment commencement to the first progression by RECIST 1.1, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse events (AEs) | Through completion of treatment, maximum 30 months
  AEs using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Objective Response Rate(ORR) | Through Study completion, until the last registered patient has been followed up for 2 years.
  ORR, defined as the proportion of patients with an objective response (CR or PR) at any stage after commencement of treatment using RECIST 1.1 criteria
Duration of response (DOR) | Through Study completion, until the last registered patient has been followed up for 2 years.
  DOR is the time between the date of first response (CR/PR per RECIST1.1) to the date of first progression per RECIST1.1. Patients who died without progression will be censored on the date of their last tumour assessment.
Overall survival (OS) | Through Study completion, until the last registered patient has been followed up for 2 years.
  OS is the time from treatment commencement to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Luen, Dr, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (4):
- Australia (4):
  - Royal North Shore, St Leonards, New South Wales
  - Mater Health, South Brisbane, Queensland
  - Monash Health, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Upon request, consideration by the Sponsor will be given to sharing reports and/or patient-level data with potential collaborators.